CLINICAL TRIAL: NCT03620097
Title: Randomized Double-blind, Parallel-group Clinical Trial, Placebo Control, to Evaluate the Efficacy and Safety of Docoxahenoic Acid in the Adjuvant Treatment of Children With Autism Spectrum Disorder.
Brief Title: Evaluate the Efficacy and Safety of DHA in the Adjuvant Treatment of Children With ASD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICI14/00355
Record Dates: First submitted 2018-07-18; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: ASD
Keywords: Autism Spectrum Disorders; ASD; Children; Autism; Docosahexaenoic acid; Inflammation; Oxidative stress; Intestinal microbiota; heavy metals
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Inflammation

STUDY DESIGN:
Intervention Model Description: The nutritional supplement used will be a product marketed according to the European Union regulation. This supplement (EUPOLY-3® DHA Infant) will be provided by Biosearch SA (Granada, Spain), as well as the placebo, in identical containers labeled with a numeric code. Product code: EUP007. The composition of both will differ only in that the formula with DHA will be fish oil refined and stabilized by the addition of soy lecithin, tocopherols of natural origin and ascorbic palmitate. In addition, its level of toxic in the raw material is controlled. This product, and the placebo, will keep the rest of the fatty acid profile similar (eg content of linoleic and linolenic fatty acids). It will be designed in a formulation suitable for preschool children with ASD; in liquid form and in a concentrated dose to ingest orally in the least amount possible (approximately 1.5cc in each dose).
Who Masked: Participant, Investigator
Masking Description: The nutritional supplement used will be a product marketed according to the European Union regulation. This supplement (EUPOLY-3® DHA Infant) will be provided by Biosearch SA (Granada, Spain), as well as the placebo, in identical containers labeled with a numeric code. Product code: EUP007. The composition of both will differ only in that the formula with DHA will be fish oil refined and stabilized by the addition of soy lecithin, tocopherols of natural origin and ascorbic palmitate. In addition, its level of toxic in the raw material is controlled. This product, and the placebo, will keep the rest of the fatty acid profile similar (eg content of linoleic and linolenic fatty acids). It will be designed in a formulation suitable for preschool children with ASD; in liquid form and in a concentrated dose to ingest orally in the least amount possible (approximately 1.5cc in each dose).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): 30 subjects will receive 800mg of DHA (Dietary Supplement: EuPoly-3 DHA Infant) per day.
  Interventions: Dietary Supplement: EuPoly-3 DHA Infant
- Control Arm (Placebo Comparator): 30 children will take a placebo with similar lipid characteristics
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: EuPoly-3 DHA Infant — Children will be selected in the first 18 months of the study, and patients with ASD will be included in the trial consecutively, and will be divided into two parallel groups according to the randomization generated by the SIGESMU® computer program with random assignment 1: 1: 30 subjects will receive 800mg of DHA per day and another 30 children, a placebo with similar lipid characteristics except that it will not have DHA content, and for a period of 6 months, double blind. After 6 months, a clinical evaluation and the same baseline analytical study will be carried out again.
  Arms: Experimental Arm
Other: Placebo — Children will be selected in the first 18 months of the study, and patients with ASD will be included in the trial consecutively, and will be divided into two parallel groups according to the randomization generated by the SIGESMU® computer program with random assignment 1: 1: 30 subjects will receive 800mg of DHA per day and another 30 children, a placebo with similar lipid characteristics except that it will not have DHA content, and for a period of 6 months, double blind. After 6 months, a clinical evaluation and the same baseline analytical study will be carried out again.
  Arms: Control Arm

SUMMARY:
In the etiopathogenesis of autistic spectrum disorder (ASD) several hypotheses have been described that include inflammation, metabolic alterations, activation of oxidative stress, changes in the intestinal microbiota and in the elimination capacity of heavy metals. Adjuvant therapies with omega-3 polyunsaturated fatty acids could modify these alterations.

DETAILED DESCRIPTION:
Several hypotheses have been described in the etiopathogenesis and evolution of ASD, among which is that there is greater oxidative stress associated with a proinflammatory state, or even metabolic alterations after exposure to heavy metals, as well as differences in intestinal microbiota. This situation could negatively influence the correct establishment of neuronal synapses and their functioning, which have still been poorly investigated, especially in children. In this way, an early intervention with nutritional supplements with DHA, which could be deficient in autism, could decrease the proinflammatory and oxidative stress state, favoring the formation of neuronal synapses as well as their activity. This intervention could positively influence to prevent the clinical deterioration associated with ASD and it would be of special interest in early childhood since at this stage of neurodevelopment there is maximum neuronal plasticity.

ELIGIBILITY:
Inclusion Criteria:

* Children and girls aged between 2 and 5 years diagnosed with Autism Spectrum Disorder according to the DSM-V criteria and the Observation Scale for the Diagnosis of Autism (ADOS).
* Informed consent signed by one of the parents or legal representative.

Exclusion Criteria:

* Children under 2 years old.
* Children diagnosed with ASD over 4 years old.
* Coexistence of another diagnosis associated with autism.
* Patients who are receiving some type of supplement or concomitant medication that does not allow a period of washing.
* Patients diagnosed with other pathologies or with mediation that may affect the study variables (oxidative stress, inflammation, cell adhesion molecules, lipid profile or microbiota).

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2015-12-02 (Actual); Study Completion 2015-12-02 (Actual)

PRIMARY OUTCOMES:
Plasma and erythrocytic level of DHA | 6 months
  Plasma and erythrocytic level of DHA in a sample of patients with ASD before and after an intervention of 6 months of treatment with 800 mg / day of DHA compared with another homogeneous group that will receive placebo.

CONTACTS AND LOCATIONS:
Overall Officials: María Mercedes Gil Campos, Doctor, Principal Investigator — Maimónides Biomedical Research Institute of Córdoba

REFERENCES:
- [Derived] de la Torre-Aguilar MJ, Gomez-Fernandez A, Flores-Rojas K, Martin-Borreguero P, Mesa MD, Perez-Navero JL, Olivares M, Gil A, Gil-Campos M. Docosahexaenoic and Eicosapentaenoic Intervention Modifies Plasma and Erythrocyte Omega-3 Fatty Acid Profiles But Not the Clinical Course of Children With Autism Spectrum Disorder: A Randomized Control Trial. Front Nutr. 2022 Mar 29;9:790250. doi: 10.3389/fnut.2022.790250. eCollection 2022. PMID 35425788